CLINICAL TRIAL: NCT01460966
Title: Assessment of Distal Protection Device in Patients at High Risk for Distal Embolism in Acute Coronary Syndrome (ACS)
Acronym: VAMPIRE3
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Yokohama City University Medical Center (Other)
Collaborators: Teikyo University (Other)
Responsible Party: Principal Investigator, Kiyoshi Hibi, Yokohama City University Medical Center, Yokohama City University Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: D110922004
Record Dates: First submitted 2011-10-17; First posted 2011-10-27 (Estimated); Last update posted 2017-04-20 (Actual); Status verified 2017-04

CONDITIONS: Coronary Artery Disease
Keywords: Distal protection device; Thrombus aspiration; Coronary Artery Disease; Coronary Disease; Acute Coronary Syndrome
MeSH Terms: conditions — Coronary Artery Disease; Coronary Disease; Acute Coronary Syndrome

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Filtrap™+ Thrombus aspiration catheter (Active Comparator)
  Interventions: Procedure: Filtrap™ + Thrombus aspiration catheter
- Thrombus aspiration catheter (Active Comparator)
  Interventions: Procedure: Thrombus aspiration catheter

INTERVENTIONS:
Procedure: Filtrap™ + Thrombus aspiration catheter — Combination of distal protection device (Filtrap™ )and thrombus aspiration catheter
  Arms: Filtrap™+ Thrombus aspiration catheter
Procedure: Thrombus aspiration catheter — Thrombus aspiration catheter only
  Arms: Thrombus aspiration catheter

SUMMARY:
Attenuated plaque ≥ 5mm by intravascular ultrasound(IVUS) was reported to be high risk for distal embolism in Acute coronary syndrome(ACS). The purpose of this study is to assess the effect of thrombus aspiration catheter and distal protection device (filter wire; Filtrap™) in the aforementioned subgroup of patients at high risk for distal embolism.

ELIGIBILITY:
Inclusion Criteria:

Patients who were diagnosed as ACS and meet the following criteria.

* Patients with acute myocardial infarction or unstable angina within 2 months from onset.
* Patients who have severe coronary stenosis which require PCI and in whom attenuated plaque ≥ 5mm (longitudinally) by IVUS before PCI is observed prior to balloon dilatation and stent deployment.

Exclusion Criteria:

* Patients who need balloon expansion (including small diameter balloon) for IVUS catheter crossing.
* Patients who were resuscitated after dead on arrival
* Graft lesion or in-stent restenosis lesion
* Patients on dialysis or renal failure (Cr>1.5mg/dl).
* Left main trunk lesion
* Target vessel size is <2.5mm or >5mm
* Ineligible for PCI
* Lactating and (possibly) pregnant woman or having possibility of pregnant
* Patients who are considered ineligible by the attending physician

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 200 (Actual)
Dates: Start 2012-07; Primary Completion 2015-12-23 (Actual); Study Completion 2017-01-31 (Actual)

PRIMARY OUTCOMES:
Incidence of no-reflow/slow-flow phenomenon after percutaneous coronary intervention (PCI) | a day

SECONDARY OUTCOMES:
Rise in CK-MB and troponin I or T the next morning after PCI (Peak of CK too in case of ST-segment elevation myocardial infarction ) | a day
Incidence of clinical events including mortality, major adverse cardiac events, and Hospitalization for heart failure | 10months
Improvement of Thrombolysis in Myocardial Infarction (TIMI) flow grade compared with baseline | 8-12months
TIMI flow grade | 8-12months
Corrected TIMI frame count | 8-12months
Myocardial blush grade | 8-12months
Incidence of any revascularization | 8-12months
Incidence of stent thrombosis | 8-12months
Plaque protrusion by IVUS inside the stent | 8-12months

CONTACTS AND LOCATIONS:
Overall Officials: Kiyoshi Hibi, Doctor, Study Chair — Yokohama City Universiy Medical Center
Locations (1):
- Yokohama City University Medical Center, Yokohama, Kanagawa, Japan

REFERENCES:
- [Derived] Hibi K, Kozuma K, Sonoda S, Endo T, Tanaka H, Kyono H, Koshida R, Ishihara T, Awata M, Kume T, Tanabe K, Morino Y, Tsukahara K, Ikari Y, Fujii K, Yamasaki M, Yamanaka T, Kimura K, Isshiki T; VAMPIRE 3 Investigators. A Randomized Study of Distal Filter Protection Versus Conventional Treatment During Percutaneous Coronary Intervention in Patients With Attenuated Plaque Identified by Intravascular Ultrasound. JACC Cardiovasc Interv. 2018 Aug 27;11(16):1545-1555. doi: 10.1016/j.jcin.2018.03.021. Epub 2018 Aug 1. PMID 30077678